CLINICAL TRIAL: NCT03012828
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Potential Effect of a Single Oral Dose of Moxidectin on the Cardiac QT Interval of Healthy Volunteers
Brief Title: Effect of a Single Oral Dose of Moxidectin on the Cardiac QT Interval of Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medicines Development for Global Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MDGH-MOX-1008
Record Dates: First submitted 2016-08-23; First posted 2017-01-06 (Estimated); Results first posted 2019-03-14 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: QT Effects in Healthy Volunteers
MeSH Terms: interventions — moxidectin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Moxidectin 4mg (Experimental): 10 subjects will receive a single oral dose of moxidectin 4mg
  Interventions: Drug: Moxidectin
- Moxidectin 8mg (Experimental): 10 subjects will receive a single oral dose of moxidectin 8mg
  Interventions: Drug: Moxidectin
- Moxidectin 16mg (Experimental): 10 subjects will receive a single oral dose of moxidectin 16mg
  Interventions: Drug: Moxidectin
- Moxidectin 24mg (Experimental): 10 subjects will receive a single oral dose of moxidectin 24mg
  Interventions: Drug: Moxidectin
- Moxidectin 36mg (Experimental): 10 subjects will receive a single oral dose of moxidectin 36mg
  Interventions: Drug: Moxidectin
- Placebo (Placebo Comparator): 10 subjects will receive a single oral dose of placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Moxidectin — Moxidectin is a broad spectrum macrocyclic lactone endectocide
  Arms: Moxidectin 16mg; Moxidectin 24mg; Moxidectin 36mg; Moxidectin 4mg; Moxidectin 8mg
Other: Placebo
  Arms: Placebo

SUMMARY:
This study will investigate the effect of a single oral dose of moxidectin on the QT interval associated with moxidectin plasma concentrations.

The effect of moxidectin on other ECG intervals, and on safety, will also be assessed, as will preliminary pharmacokinetics and metabolism

DETAILED DESCRIPTION:
Moxidectin is being developed as a treatment for Onchocerciasis (river blindness), a serious, debilitating, disease caused by a parasitic worm, Onchocerca volvulus.

Five dose levels of moxidectin will be administered to healthy volunteers and ECG assessments undertaken at pre-specified pharmacokinetic time points to correlate QT interval with moxidectin concentration in plasma.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male between 18 and 50 years of age (inclusive);
2. Body mass index (BMI) of 18 to 30 kg/m2 (inclusive) and a minimum weight of 50 kg (110 lbs);
3. Biologically or surgically sterile or must commit to using a reliable method of birth control, in the opinion of the investigator, from Screening through the duration of the study;
4. Willing and able to give written informed consent.

Exclusion Criteria:

1. Unwilling to abstain from alcohol, caffeine, xanthine containing products, Seville oranges, grapefruit juices, and fish liver oils within 72 hours before Check in (Day -1) and throughout the inpatient period of the study;
2. Less than 1 bowel movement every 24 hours in the absence of any laxative, suppository, or enema use during the month before Screening;
3. Abnormal fecal consistency within 24 hours of Check in (Day -1);
4. Clinically relevant abnormal findings on medical history, clinical laboratory test results, vital sign measurements, safety 12 lead ECG results, or physical examination at Screening or Baseline which, in the opinion of the investigator, would interfere with dosing, jeopardize the safety of the subject, or impact the validity of the study results;
5. History of clinically significant dermatologic, gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, psychiatric, or cardiovascular disease or any other condition which, in the opinion of the investigator, would interfere with dosing, jeopardizes the safety of the subject, or impacts the validity of the study results;
6. History or hypersensitivity or allergic reactions to ivermectin, moxidectin, or any of the ingredients in the study drug as described in the Investigator's Brochure;
7. Any condition that may affect oral drug absorption (eg, previous surgery on the gastrointestinal tract including removal of parts of the stomach, bowel, liver, gall bladder, or pancreas);
8. History of risk factors for torsades de pointes, including unexplained syncope, known long QT syndrome, heart failure, myocardial infarction, angina, or clinically significant abnormal laboratory assessments including hypokalemia, hypercalcemia, or hypomagnesemia. Subjects are also excluded if there is a family history of long QT syndrome or Brugada syndrome;
9. A sustained supine systolic blood pressure >150 mm Hg or <90 mm Hg or a supine diastolic blood pressure >95 mm Hg or <50 mm Hg at Screening or Check in (Day -1). Blood pressure may be retested twice in the supine position. The blood pressure abnormality is considered sustained if either the systolic or the diastolic blood pressure values are outside of the stated limits after 3 assessments, and the subject will not to be randomized;
10. A resting heart rate (HR) of <40 beats per minute (bpm) or >100 bpm when vital signs are measured at Screening or Check in (Day -1);
11. An uninterpretable or abnormal screening ECG indicating a second or third degree atrioventricular block, or 1 or more of the following: QRS interval >110 milliseconds (msec); QT interval corrected by Fridericia's formula (QTcF) >450 msec; PR interval >200 msec; or any rhythm other than sinus rhythm that is interpreted by the investigator to be clinically significant;
12. Concomitant use of prescription medications, including medications known to prolong the corrected QT interval (QTc) or herbal preparations, within 14 days or 5 half-lives (whichever is longer) before study drug dosing, or use of an over the counter (OTC) medication or vitamins within 7 days before study drug dosing;
13. Received an investigational drug during the 30 days, or 5 half lives of the study drug (whichever is longer), before Check in (Day -1) or is planning to receive another investigational drug at any time during the study;
14. History or presence of alcohol abuse (defined as consumption of more than 210 mL of alcohol per week, or the equivalent of fourteen 4 ounce [oz] glasses of wine or fourteen 12 oz cans/bottles of beer or wine coolers per week) within 6 months before Screening or positive alcohol test at Screening or Check-in (Day -1);
15. History or presence of substance abuse within the past 2 years or positive drug screen test at Screening or Check in (Day -1);
16. Current use or has used tobacco- or nicotine-containing products (eg, cigarettes, cigars, chewing tobacco, snuff, etc.) within 14 days before study drug dosing;
17. Blood donation or significant blood loss within 30 days before Check-in (Day -1) or donated plasma within 7 days before Check-in (Day -1);
18. Presence of hepatitis B surface antigen or antibodies to human immunodeficiency virus (HIV) or hepatitis C virus at Screening;
19. Poor venous access in both arms;
20. Unable to understand verbal or written English or any other language for which a certified translation of the informed consent form is available;
21. For any reason, is deemed by the investigator or medically qualified designee to be inappropriate for this study, including a subject who is unable to communicate or cooperate with the investigator, and/or is unwilling to comply with protocol defined procedures and complete the study.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-01; Primary Completion 2017-03 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Sullivan, Study Director — Sponsor GmbH
Locations (1):
- Spaulding Clinical, West Bend, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
Healthy volunteer study: results are not useful to individuals

REFERENCES:
- [Derived] Kinrade SA, Mason JW, Sanabria CR, Rayner CR, Bullock JM, Stanworth SH, Sullivan MT. Evaluation of the Cardiac Safety of Long-Acting Endectocide Moxidectin in a Randomized Concentration-QT Study. Clin Transl Sci. 2018 Nov;11(6):582-589. doi: 10.1111/cts.12583. Epub 2018 Sep 19. PMID 30117300

RESULTS

PARTICIPANT FLOW:
Groups:
- Moxidectin 4mg: 10 subjects will receive a single oral dose of moxidectin 4mg
  Moxidectin
- Moxidectin 8mg: 10 subjects will receive a single oral dose of moxidectin 8mg
  Moxidectin
- Moxidectin 16mg: 10 subjects will receive a single oral dose of moxidectin 16mg
  Moxidectin
- Moxidectin 24mg: 10 subjects will receive a single oral dose of moxidectin 24mg
  Moxidectin
- Moxidectin 36mg: 10 subjects will receive a single oral dose of moxidectin 36mg
  Moxidectin
- Placebo: 10 subjects will receive a single oral dose of placebo
  Placebo
Period: Overall Study
Arm/Group | Moxidectin 4mg | Moxidectin 8mg | Moxidectin 16mg | Moxidectin 24mg | Moxidectin 36mg | Placebo
Started | 10 | 10 | 10 | 10 | 10 | 10
Completed | 9 | 10 | 8 | 10 | 8 | 8
Not Completed | 1 | 0 | 2 | 0 | 2 | 2
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Non-compliance with protocol | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Delay to last visit would delay DBL | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Moxidectin 4mg | Moxidectin 8mg | Moxidectin 16mg | Moxidectin 24mg | Moxidectin 36mg | Placebo | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.1 (7.77) | 30.4 (8.73) | 30.9 (8.32) | 31.2 (8.27) | 30.2 (8.87) | 32.3 (6.72) | 32.0 (8.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 10 | 10 | 10 | 10 | 10 | 10 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 1 | 1 | 0 | 0 | 6
  Not Hispanic or Latino | 8 | 8 | 9 | 9 | 10 | 10 | 54
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Black or African American | 3 | 7 | 4 | 5 | 5 | 5 | 29
  White | 7 | 3 | 5 | 4 | 3 | 5 | 27
  More than one race | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 10 | 10 | 10 | 60
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram /meter squared (kg/m2)] | 26.2 (3.74) | 24.9 (3.35) | 25.8 (3.71) | 25.1 (3.00) | 26.7 (3.09) | 26.1 (3.11) | 25.8 (3.26)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in QTc Interval (Corrected by Friderica's Formula, dQTcF) Associated With Plasma Moxidectin Concentrations After a Single Dose
Description: Triplicate 10-second ECG recordings taken 1 minute apart using a Mortara continuous 12-lead digital ECG recorder connected to each subject during the Baseline to 72-hour post dose confinement period. Baseline only and baseline and placebo adjusted changes in QTc interval (corrected using the Friderica formula, QTcF) at each timepoint for each dose level were determined. The mean change from baseline (without and with placebo correction, dQTcF and ddQTcF respectively) at each of the 14 time points was calculated for each dose level. The primary outcome measure was the mean dQTcF for all subjects(the dQTcF gradient). The mean dQTcF for each active treatment group was determined at each post dose timepoint but the mean dQTcF by dose level was not calculated. The mean dQTcF at approximate moxidectin Tmax (hour 3 or hour 4) for each active treatment group and at hour 3 for the placebo group is reported.
Time Frame: Baseline (pre-dose) and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 60, and 72 hours post dosing
Population: The ECG population included all subjects who received one dose of study drug and have at least 1 pair of pre-dose and post-dose QTc interval and was used in the model.
Measure: Mean (90% Confidence Interval); unit: millseconds
Groups:
- All Subjects: 50 subjects received a single dose of between 4mg and 36mg of moxidectin. 10 subjects received a dose of placebo,
Arm/Group | Moxidectin 4mg | Moxidectin 8mg | Moxidectin 16mg | Moxidectin 24mg | Moxidectin 36mg | Placebo | All Subjects
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 60
millseconds | -5.1 [-10.90 to 0.68] | -4.5 [-9.19 to 0.27] | -4.5 [-8.39 to -0.63] | -6.3 [-12.68 to 0.04] | -3.9 [-7.77 to 0.03] | -2.9 [-6.58 to 0.76] | -0.0077 [-0.0255 to 0.0101]
Statistical Analysis 1: Comparison: All Subjects; The primary analysis used a mixed-effects model to explore the relationship between the time-matched, baseline-adjusted QTcF (delta (d)QTcF) and moxidectin concentrations. dQTcF was a dependent variable and treatment, time point, and treatment by time point interaction as the independent variables with baseline QTcF as a covariate and time-matched concentrations of moxidectin as a covariate with random effects of intercept and slope for each subject.Concentrations of zero were used for placebo; Test type: Other — The model was used for predicting population average and 90% 2-sided bootstrapped CI of the baseline-adjusted difference between active and placebo at each time point bound at clinically relevant concentrations; p = 0.4727, Mixed Models Analysis; Slope = -0.0077, 90% CI 2-sided [-0.0255 to 0.0101] — The primary mixed effects model analysis revealed a nearly flat dQTcF - plasma concentration gradient

2. Secondary Outcome: Concentrations of Moxidectin in Plasma
Description: Concentrations of moxidectin in plasma were assessed by collection of plasma samples at pre-specified intervals after oral dosing with moxidectin. The concentration of moxidectin was determined using a validated LC MS/MS method.The pharmacokinetic time points coincided with ECG collection timepoints (within 5 minutes and no later than 10 minutes after ECG recordings). Plasma PK parameters were estimated from the concentration measurements, including maximum concentration (Cmax) for each individual and mean for each dose cohort.
Time Frame: Pre-dose and at 0.5, 1, 2, 3, 4, 5, 6, 8, 12*, 24, 36, 48, 60, and 72 hours and days 8,15 and 22 post dosing
Population: Pharmacokinetic population - includes all subjects who received at least 1 dose of moxidectin and provide an adequate number of plasma samples for determination of PK parameters, analyzed according to drug received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter
Arm/Group | Moxidectin 4mg | Moxidectin 8mg | Moxidectin 16mg | Moxidectin 24mg | Moxidectin 36mg
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
nanogram/milliliter | 27.2 (30.6) | 56.7 (20.8) | 133 (27.1) | 176 (18.7) | 247 (19.7)

3. Other Pre Specified Outcome: Subjects With Categorical Changes From Baseline in 12-lead Electrocardiograms (ECGs)
Description: Changes from baseline in QTcF exceeding regulatory standard categorical limits (> 30msec change or exceeding 450msec). Report applies to changes of 30msec - </= 60msec only
Time Frame: At Baseline and Days 1, 2, 3, 4, 22 and Week 12
Population: Safety population - all who received at least one dose of study drug
Measure: Number; unit: participants
Arm/Group | Moxidectin 4mg | Moxidectin 8mg | Moxidectin 16mg | Moxidectin 24mg | Moxidectin 36mg | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10
participants | 1 | 0 | 0 | 0 | 1 | 1

4. Other Pre Specified Outcome: Change From Baseline in Heart Rate (HR) and Duration of Other Interval Parameters (PR and QRS)
Description: Changes from Baseline were assessed at each timepoint up to 72 hours post dose. Mean changes across the 72 hour assessment period for each parameter were calculated for each moxidectin group and the placebo group and for the population overall.
Time Frame: Baseline (pre-dose) and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 60, and 72 hours post dosing
Population: ECG population - all subjects who receive one dose of study drug and have at least one pair of pre-dose and post-dose QTc data, analyzed as randomized
Measure: Mean (95% Confidence Interval); unit: milliseconds
Groups:
- All Subjects: 50 subjects received a single dose of moxidectin between 4mg and 36mg and 10 subjects received placebo
Arm/Group | Moxidectin 4mg | Moxidectin 8mg | Moxidectin 16mg | Moxidectin 24mg | Moxidectin 36mg | Placebo | All Subjects
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 60
milliseconds
  Change in Heart rate (HR) | -1.0 [-4.80 to 2.76] | 0.5 [-2.79 to 3.85] | -1.1 [-6.35 to 4.07] | -3.6 [-10.93 to 3.65] | -1.5 [-7.34 to 4.42] | -2.9 [-6.21 to 0.39] | -0.005 [-0.018 to 0.009]
  Change in PR interval | 2.2 [-0.49 to 4.87] | -0.1 [-5.84 to 5.66] | -2.1 [-7.63 to 3.47] | 4.6 [-3.10 to 12.34] | -3.5 [-8.86 to 1.92] | -1.8 [-5.64 to 1.98] | -0.002 [-0.016 to 0.012]
  Change in QRS interval | -1.6 [-3.26 to 0.10] | -0.7 [-5.38 to 3.94] | 0.4 [-1.75 to 2.49] | -0.8 [-3.55 to 2.03] | 0.4 [-2.00 to 2.86] | 1.2 [-0.29 to 2.59] | 0.004 [-0.003 to 0.012]

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the full 12 weeks of study follow-up
Arm/Group | Moxidectin 4mg | Moxidectin 8mg | Moxidectin 16mg | Moxidectin 24mg | Moxidectin 36mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 3/10 | 3/10 | 1/10 | 0/10 | 3/10 | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Moxidectin 4mg (N=10) | Moxidectin 8mg (N=10) | Moxidectin 16mg (N=10) | Moxidectin 24mg (N=10) | Moxidectin 36mg (N=10) | Placebo (N=10)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Medical device site reaction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
AST increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood cholesterol increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-03-01): https://cdn.clinicaltrials.gov/large-docs/28/NCT03012828/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-01): https://cdn.clinicaltrials.gov/large-docs/28/NCT03012828/SAP_001.pdf